CLINICAL TRIAL: NCT02223273
Title: A Cluster Randomized Trial to Evaluate the Increase in Usage of Evidence-based Practices for Stroke Treatment Using a Multifaceted Strategy
Brief Title: Brazilian Intervention to Increase Evidence Usage in Practice - Stroke (BRIDGE-Stroke)
Acronym: BRIDGEStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BRIDGE-Stroke
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke,; quality improvement
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifaceted Strategy (Experimental): Multifaceted Intervention
  1. Simulation Based Team Training
  2. Case Manager
  3. Check lists
  4. Reminders
  5. Educational Materials
  Interventions: Behavioral: Multifaceted Strategy
- Usual Care (No Intervention): Hospital Standard Treatment

INTERVENTIONS:
Behavioral: Multifaceted Strategy — 1. Simulation Based Team Training
  2. Case Manager: a trained person who works in the hospital and is responsible for ensuring the usage of all interventions
  3. Reminders -
  4. Check lists - decision support algorithm
  5. Distribution of educational materials: guidelines and recommendations for best practices
  Arms: Multifaceted Strategy

SUMMARY:
Phase 1: An observational study ( registry) will be conducted with the objective of documenting the practice of stroke treatment in brazilian and latin american hospitals.

Phase 2: A cluster randomized trial aiming to evaluate the effect of a multifaceted strategy to increase evidence based treatments usage for stroke patients. The hospitals will be randomized into two groups: the multifaceted strategy group and the usual care group.

DETAILED DESCRIPTION:
Study Objective: The purpose of this study is to evaluate a multifaceted strategy to increase evidence based therapies for patients with acute ischemic stroke.

Study Population; Patients with suspected stroke or transient ischemic attack (TIA) with symptoms lasting up to 24h hours.

Quality Improvement Multifaceted Intervention: The strategy includes a simulation based team training, case manager, check lists, reminders and educational material.

ELIGIBILITY:
Patient Eligibility Criteria

Inclusion Criteria:

* Patients over 18 years old, diagnosed with ischemic stroke (including transient ischemic attack) with symptoms lasting up to 24 hours.

Exclusion Criteria:

* Patients with signs of hemorrhagic stroke, expansive lesions, central nervous system infections, and those coming from institutions that did not provide institutional approval form signed by the patients' guardians.

Cluster Eligibility Criteria

Inclusion Criteria:

* Hospitals with a emergency department, with available tomography, neurologist and alteplase

Exclusion Criteria:

* Hospitals that don't provide Institutional Authorization Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1624 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Frequency of Evidence Based Strategies | Discharge or 7 days after admission
  For phase 1: Proportion of prescription of evidence-based strategies. in the first 48 hours and prior to discharge
Composite Adherence Score | Discharge or 7 days after admission
  Composite Adherence Score: defined as the sum of usage of evidence based therapies in the first 48 hours and at discharge among the patients' total eligible opportunities. For this purpose, patients with contraindications (which are specific for each endpoint) were excluded from the denominators. Evidence based therapies in the first 48 hours include: antithrombotics within 48 hours of admission, use of recombinant Plasminogen Activator (Rt-PA)in patients who arrive at the hospital within 3.5 hours of symptom onset and who are treated within 4.5 hours of symptom onset, dysphagia screening, pre-deep venous thrombosis prophylaxis, door to needle time < 60 minutes, dysphagia screening). Discharge Therapies include: antithrombotics, lipid lowering agents in patients with LDL 100 or not documented, anticoagulants for atrial fibrilation or flutter, assessment for rehabilitation and smoke cessation education

SECONDARY OUTCOMES:
"All or None" Quality Measures | Discharge or 7 days after admission
  Proportion of prescription of evidence-based strategies in the first 48 hours and at discharge "All or none" measures including the evidence based therapies in the first 48h: antithrombotics, use of recombinant Plasminogen Activator (Rt-PA)in patients who arrive at the hospital within 3.5 hours of symptom onset and who are treated within 4.5 hours of symptom onset, dysphagia screening, pre-deep venous thrombosis prophylaxis, door to needle time < 60 minutes, dysphagia screening). Discharge Therapies include: antithrombotics, lipid lowering agents in patients with LDL 100 or not documented, anticoagulants for atrial fibrilation or flutter, assessment for rehabilitation and smoke cessation education
Additional Strategies | Discharge or 7 days after admission
  Proportion of usage of the additional strategies: use of recombinant Plasminogen Activator (Rt-PA), anti-hypertensive agents, and door to needle time< 45 min)
Total Mortality | Discharge or 7 days after admission and 90 days
  In hospital and 90 days mortality
Disability | 90 days
  Degree of disability (measured by the Modified Rankin Scale) at discharge and in 90 days.
Stroke Recurrence | 90 days
  Number of patients presenting a new stroke in 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, MD, PhD, Study Chair — Hospital do Coração; M. Julia Machline Carrion, MD, MHS, PhD, Principal Investigator — Hospital do Coração
Locations (1):
- Brazil, São Paulo, Brazil

REFERENCES:
- [Derived] Machline-Carrion MJ, Santucci EV, Damiani LP, Bahit MC, Malaga G, Pontes-Neto OM, Martins SCO, Zetola VF, Normilio-Silva K, Rodrigues de Freitas G, Gorgulho A, De Salles A, Pacheco da Silva BG, Santos JY, de Andrade Jesuino I, Bueno PRT, Cavalcanti AB, Guimaraes HP, Xian Y, Bettger JP, Lopes RD, Peterson ED, Berwanger O; BRIDGE-Stroke Investigators. Effect of a Quality Improvement Intervention on Adherence to Therapies for Patients With Acute Ischemic Stroke and Transient Ischemic Attack: A Cluster Randomized Clinical Trial. JAMA Neurol. 2019 Aug 1;76(8):932-941. doi: 10.1001/jamaneurol.2019.1012. PMID 31058947
- [Derived] Machline-Carrion MJ, Santucci EV, Damiani LP, Bahit C, Malaga G, Pontes-Neto OM, Martins SCO, Zetola VF, Normilio-Silva K, de Freitas GR, Gorgulho A, De Salles A, da Silva BGP, Santos JY, de Andrade Jesuino I, Bueno PRT, Cavalcanti AB, Guimaraes HP, Xian Y, Bettger JP, Lopes RD, Peterson ED, Berwanger O. An international cluster-randomized quality improvement trial to increase the adherence to evidence-based therapies for acute ischemic stroke and transient ischemic attack patients: Rationale and design of the BRIDGE STROKE Trial. Am Heart J. 2019 Jan;207:49-57. doi: 10.1016/j.ahj.2018.09.009. Epub 2018 Sep 30. PMID 30415083